CLINICAL TRIAL: NCT00095498
Title: A Randomized, Double-blind, Placebo-controlled, Multi-dose Phase 2 Study to Determine the Efficacy, Safety and Tolerability of Denosumab in the Treatment of Rheumatoid Arthritis
Brief Title: Efficacy, Safety and Tolerability of Denosumab in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20040144
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
Keywords: arthritis; joint pain; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Arthralgia | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Denosumab 180 mg (Experimental): Participants received 180 mg denosumab by subcutaneous injection on Day 1 and at Month 6.
  Interventions: Drug: denosumab
- Denosumab 60 mg (Experimental): Participants received 60 mg denosumab by subcutaneous injection on Day 1 and at Month 6.
  Interventions: Drug: denosumab
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections on Day 1 and at Month 6.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo subcutaneous injection
  Arms: Placebo
Drug: denosumab — For subcutaneous injection
  Other Names: AMG 162
  Arms: Denosumab 180 mg; Denosumab 60 mg

SUMMARY:
This study will determine the efficacy, safety, and tolerability of denosumab (AMG 162) in the treatment of Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA.
* All subjects will be required to have been taking a stable dose of methotrexate.
* Active RA at screening defined as greater than or equal to 6 swollen joints.
* The presence of erosive disease

Exclusion Criteria:

* Received any biologic agent (e.g., Enbrel®, Remicade®, Humira®, Kineret®) or Arava® within 8 weeks before randomization; past use of these agents is allowed.
* Steroid use greater than 15 mg/day.
* Scheduled for surgery or joint replacement in the hands, wrists or feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2004-08-11 (Actual); Primary Completion 2007-04-01 (Actual); Study Completion 2007-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cohen SB, Dore RK, Lane NE, Ory PA, Peterfy CG, Sharp JT, van der Heijde D, Zhou L, Tsuji W, Newmark R; Denosumab Rheumatoid Arthritis Study Group. Denosumab treatment effects on structural damage, bone mineral density, and bone turnover in rheumatoid arthritis: a twelve-month, multicenter, randomized, double-blind, placebo-controlled, phase II clinical trial. Arthritis Rheum. 2008 May;58(5):1299-309. doi: 10.1002/art.23417. PMID 18438830
- [Background] Deodhar A, Dore RK, Mandel D, Schechtman J, Shergy W, Trapp R, Ory PA, Peterfy CG, Fuerst T, Wang H, Zhou L, Tsuji W, Newmark R. Denosumab-mediated increase in hand bone mineral density associated with decreased progression of bone erosion in rheumatoid arthritis patients. Arthritis Care Res (Hoboken). 2010 Apr;62(4):569-74. doi: 10.1002/acr.20004. PMID 20391513
- [Background] Dore RK, Cohen SB, Lane NE, Palmer W, Shergy W, Zhou L, Wang H, Tsuji W, Newmark R; Denosumab RA Study Group. Effects of denosumab on bone mineral density and bone turnover in patients with rheumatoid arthritis receiving concurrent glucocorticoids or bisphosphonates. Ann Rheum Dis. 2010 May;69(5):872-5. doi: 10.1136/ard.2009.112920. Epub 2009 Sep 3. PMID 19734132
- [Background] Sharp JT, Tsuji W, Ory P, Harper-Barek C, Wang H, Newmark R. Denosumab prevents metacarpal shaft cortical bone loss in patients with erosive rheumatoid arthritis. Arthritis Care Res (Hoboken). 2010 Apr;62(4):537-44. doi: 10.1002/acr.20172. PMID 20391509
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_49_AMG_162_20040144.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 11-Aug-2004 Last Subject Enrolled: 07-Apr-2005
Period: Overall Study
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Started | 76 | 73 | 78
Received Investigational Product | 72 | 71 | 75
Completed | 39 | 38 | 39
Not Completed | 37 | 35 | 39
Not completed — Physician Decision | 9 | 10 | 8
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 16 | 15
Not completed — Disease progression | 0 | 1 | 1
Not completed — Ineligibility determined | 3 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Noncompliance | 1 | 0 | 1
Not completed — Other | 6 | 7 | 6
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Requirement for alternative therapy | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo | Total
Number analyzed (Participants) | 76 | 73 | 78 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (11) | 57.3 (11.4) | 57 (11.1) | 57.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 62 | 166
  Male | 23 | 22 | 16 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2 | 4
  Japanese | 1 | 0 | 1 | 2
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  White or Caucasian | 66 | 59 | 62 | 187
  Black or African American | 1 | 3 | 2 | 6
  Hispanic or Latino | 6 | 6 | 9 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Other | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Rheumatoid Arthritis Erosion Score Measured From MRI Assessments (RA-MRI ES) at Month 6
Description: Fifteen sites in each wrist and 10 sites in each hand were assessed by a blinded and independent reader. Each site was scored from 0 to 10 (in accordance with the European League Against Rheumatism [EULAR]-Outcome Measures in Rheumatology Clinical Trials convention), with each unit increment representing 10% incremental loss of the peripheral 1 cm of articular bone. The Erosion Score is a sum of erosion scores from 50 joint sites in both hands/wrists and ranges from 0 (normal, no erosion) to 500 (worst possible erosion).
Time Frame: Baseline, Month 6
Population: All randomized patients who received at least 1 dose of investigational product with a non-missing baseline and at least 1 non-missing postbaseline measurement, and with available data at 6 months.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 67 | 66
units on a scale | 0.00 (3.49) [-13.00 to 12.53] | 0.00 (3.43) [-17.86 to 9.00] | 0.49 (5.08) [-5.50 to 37.00]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.264, van Elteren stratified rank test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.018, van Elteren stratified rank test

2. Secondary Outcome: Change From Baseline in Radiographic Total Modified Sharp Score (TSS) at Month 12
Description: TSS is the sum of erosion and joint space narrowing scores obtained from radiographs of the hands and feet, assessed by 2 independent readers. The joint erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints in the feet. Each joint was scored, according to the surface area involved, from 0 (no erosion) to 5 (extensive loss of bone from more than one half of the articulating bone). Because each side of a foot joint was graded on this scale, the maximum erosion score for a foot joint was 10 and the maximal erosion score was 280. Joint Space Narrowing (JSN) Score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet. Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, was scored from 0 (normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. The TSS ranged from 0 (normal) to 448 (worst).
Time Frame: Baseline, Month 12
Population: All randomized patients who received at least 1 dose of investigational product with a non-missing baseline and at least 1 non-missing postbaseline measurement, and with available data at 12 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 71
units on a scale | 0 [0 to 1.5] | 0 [-0.5 to 1] | 0.5 [0 to 2]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.032, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.180, van Elteren Stratified Rank Test

3. Secondary Outcome: Change From Baseline in Radiographic Total Modified Sharp Score (TSS) at Month 6
Description: as for outcome 2
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 69 | 71
units on a scale | 0 [0 to 0.5] | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.602, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.181, van Elteren Stratified Rank Test

4. Secondary Outcome: Change From Baseline in Radiographic Erosion Score at Month 12
Description: The joint erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints in the feet, obtained from radiographs of the hands and feet and assessed by 2 independent readers. Each joint was scored, according to the surface area involved, from 0 (no erosion) to 5 (extensive loss of bone from more than one half of the articulating bone). Because each side of a foot joint was graded on this scale, the maximum erosion score for a foot joint was 10 and the maximal erosion score was 280.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 71
units on a scale | 0 [0 to 0.5] | 0 [0 to 0.5] | 0 [0 to 1.5]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.012, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.007, van Elteren Stratified Rank Test

5. Secondary Outcome: Change From Baseline in Radiographic Erosion Score at Month 6
Description: as for outcome 4
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 69 | 71
units on a scale | 0 [0 to 0] | 0 [0 to 0.5] | 0 [0 to 0.5]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.277, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.019, van Elteren Stratified Rank Test

6. Secondary Outcome: Change From Baseline in Radiographic Joint Space Narrowing Score at Month 12
Description: Joint Space Narrowing (JSN) Score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet obtained from radiographs of the hands and feet and assessed by 2 independent readers. Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, was scored from 0 (normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score (indicating worst joint space narrowing) of 168.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 71
units on a scale | 0 [0 to 1] | 0 [0 to 0.5] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.382, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.488, van Elteren Stratified Rank Test

7. Secondary Outcome: Change From Baseline in Radiographic Joint Space Narrowing Score at Month 6
Description: as for outcome 6
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 69 | 71
units on a scale | 0 [0 to 0.5] | 0 [0 to 0.97] | 0 [0 to 0.5]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.236, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.712, van Elteren Stratified Rank Test

8. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 1
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from baseline to Month 1 calculated using ((month 1 value - baseline value) / baseline value ) x 100. Least squares means are based on a repeated measures model adjusting for treatment, visit, baseline value, and strata (4 strata from the combination of baseline use of steroid and previous use of biologic).
Time Frame: Baseline, Month 1
Population: All randomized patients who received at least 1 dose of investigational product with a non-missing baseline and at least 1 non-missing postbaseline measurement, and with available data at 1 month.
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 66 | 66
Percent change from baseline | 0.25 (0.29) | 0.59 (0.29) | -0.34 (0.29)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.026, Repeated Measures Model; Mean Difference (Final Values) = 0.93, 95% CI [0.11 to 1.74]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.155, Repeated measures model; Mean Difference (Final Values) = 0.59, 95% CI [-0.23 to 1.41]

9. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 6
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from baseline to month 6 calculated using ((month 6 value - baseline value) / baseline value ) x 100. Least squares means are based on a repeated measures model adjusting for treatment, visit, baseline value, and strata (4 strata from the combination of baseline use of steroid and previous use of biologic).
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 68
Percent change from baseline | 2.61 (0.38) | 2.40 (0.37) | 0.73 (0.38)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Repeated Measures Model; Mean Difference (Final Values) = 1.67, 95% CI [0.62 to 2.72]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 1.89, 95% CI [0.84 to 2.94]

10. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from baseline to Month 12 calculated using ((Month 12 value - baseline value) / baseline value ) x 100. Least squares means based on repeated measures model adjusting for treatment, visit, baseline value, and strata (4 strata from the combination of baseline use of steroid and previous use of biologic).
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 62 | 66 | 62
Percent change from baseline | 4.09 (0.40) | 3.00 (0.39) | 0.80 (0.40)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 2.2, 95% CI [1.1 to 3.29]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 3.29, 95% CI [2.18 to 4.39]

11. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density at Month 1
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from baseline to Month 1 calculated using ((Month 1 value - baseline value) / baseline value ) x 100.
  Least squares means based on repeated measures model adjusting for treatment, visit, baseline value, and strata (4 strata from the combination of baseline use of steroid and previous use of biologic).
Time Frame: Baseline, Month 1
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 65
Percent change from baseline | 0.64 (0.38) | -0.15 (0.38) | -0.16 (0.38)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.986, Repeated Measures Model; Mean Difference (Final Values) = 0.01, 95% CI [-1.06 to 1.08]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.141, Repeated Measures Model; Mean Difference (Final Values) = 0.8, 95% CI [-0.27 to 1.86]

12. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density at Month 6
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from baseline to Month 6 calculated using ((Month 6 value - baseline value) / baseline value ) x 100. Least squares means based on repeated measures model adjusting for treatment, visit, baseline value, and strata (4 strata from the combination of baseline use of steroid and previous use of biologic).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 68 | 69
Percent change from baseline | 0.84 (0.37) | 0.89 (0.37) | -0.06 (0.37)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.073, Repeated Measures Model; Mean Difference (Final Values) = 0.95, 95% CI [-0.09 to 1.99]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.09, Repeated Measures Model; Mean Difference (Final Values) = 0.89, 95% CI [-0.14 to 1.93]

13. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density at Month 12
Description: as for outcome 10
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 63
Percent change from baseline | 1.51 (0.47) | 1.34 (0.47) | -0.47 (0.47)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.007, Repeated Measures Model; Mean Difference (Final Values) = 1.81, 95% CI [0.51 to 3.12]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.003, Repeated Measures Model; Mean Difference (Final Values) = 1.98, 95% CI [0.67 to 3.29]

14. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density at Month 1
Description: as for outcome 11
Time Frame: Baseline, Month 1
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 65
Percent change from baseline | 0.06 (0.22) | 0.00 (0.22) | -0.02 (0.22)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.938, Repeated Measures Model; Mean Difference (Final Values) = 0.02, 95% CI [-0.58 to 0.63]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.787, Repeated Measures Model; Mean Difference (Final Values) = 0.08, 95% CI [-0.53 to 0.69]

15. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density at Month 6
Description: as for outcome 12
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 68 | 69
Percent change from baseline | 1.12 (0.24) | 0.95 (0.24) | -0.06 (0.24)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Repeated Measures Model; Mean Difference (Final Values) = 1, 95% CI [0.33 to 1.67]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 1.18, 95% CI [0.51 to 1.85]

16. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density at Month 12
Description: as for outcome 10
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 63
Percent change from baseline | 1.67 (0.33) | 1.56 (0.33) | -0.38 (0.33)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 1.94, 95% CI [1.02 to 2.85]
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Model; Mean Difference (Final Values) = 2.04, 95% CI [1.13 to 2.96]

17. Secondary Outcome: Percent Change From Baseline in Serum Collagen C-Telopeptide (CTX) at Month 3
Description: Percent change from baseline to Month 3 in serum Collagen C-Telopeptide (CTX) Type I calculated using ((Month 3 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 3
Population: All randomized patients who received at least 1 dose of investigational product with a non-missing baseline and at least 1 non-missing postbaseline measurement, and with available data at 3 months.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 69
Percent change from baseline | -78.67 [-86.29 to -62.86] | -80.46 [-86.27 to -66.84] | -11.48 [-26.95 to 15.59]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

18. Secondary Outcome: Percent Change From Baseline in Serum CTX at Month 6
Description: Percent change from baseline to Month 6 in serum Collagen C-Telopeptide (CTX) Type I calculated using ((Month 6 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 68 | 67
Percent change from baseline | -62.69 [-78.56 to -46.23] | -50.64 [-63.31 to -22.37] | -12.94 [-31.20 to 23.30]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

19. Secondary Outcome: Percent Change From Baseline in Serum CTX at Month 12
Description: Percent change from Baseline to Month 12 in serum C-Telopeptide (CTX) Type I calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 62 | 66 | 62
Percent change from baseline | -65.65 [-78.62 to -48.40] | -47.24 [-63.60 to -27.20] | -23.36 [-45.43 to 1.67]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

20. Secondary Outcome: Percent Change From Baseline in Procollagen 1 N-terminal Peptide (P1NP) at Month 3
Description: Percent change from baseline to Month 3 in procollagen 1 N-terminal peptide (P1NP) calculated using ((Month 3 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 3
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 69
Percent change from baseline | -55.08 [-69.30 to -44.40] | -57.57 [-70.07 to -46.07] | -12.23 [-21.57 to -0.11]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

21. Secondary Outcome: Percent Change From Baseline in P1NP at Month 6
Description: Percent change from baseline to Month 6 in procollagen 1 N-terminal peptide (P1NP) calculated using ((Month 6 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 68 | 67
Percent change from baseline | -57.06 [-67.17 to -37.13] | -51.57 [-64.51 to -37.35] | -22.17 [-39.69 to -3.07]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

22. Secondary Outcome: Percent Change From Baseline in P1NP at Month 12
Description: Percent change from baseline to Month 12 in procollagen 1 N-terminal peptide (P1NP) calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 33 | 39 | 30
Percent change from baseline | -45.84 [-61.36 to -30.09] | -41.8 [-57.30 to -18.89] | -17.53 [-31.42 to -0.02]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.016, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

23. Secondary Outcome: Percent Change From Baseline in Urine Type II Collagen C-telopeptide (C-Tx) /Creatinine at Month 3
Description: Percent change from baseline to Month 3 in urine Type II collagen C-Telopeptide (CTX)/Creatinine calculated using ((Month 3 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 3
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 63 | 65
Percent change from baseline | -46.59 [-71.58 to 4.17] | -35.8 [-56.80 to 16.99] | 2.71 [-24.18 to 31.72]
Statistical Analysis 1: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, van Elteren Stratified Rank Test

24. Secondary Outcome: Percent Change From Baseline in Urine Type II C-Tx /Creatinine at Month 6
Description: Percent change from baseline to Month 6 in urine Type II collagen C-Telopeptide (CTX)/Creatinine calculated using ((Month 6 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 56 | 63 | 63
Percent change from baseline | 7.17 [-32.43 to 88.27] | 9.65 [-21.79 to 51.16] | 4.54 [-27.44 to 56.52]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.673, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.589, van Elteren Stratified Rank Test

25. Secondary Outcome: Percent Change From Baseline in Urine Type II C-Tx /Creatinine at Month 12
Description: Percent change from baseline to Month 12 in urine Type II collagen C-Telopeptide (CTX)/Creatinine calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 29 | 35 | 22
Percent change from baseline | 36.92 [4.50 to 111.51] | 61.92 [-15.84 to 108.60] | -3.93 [-37.70 to 126.65]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.175, van Elteren Stratified Rank Test
Statistical Analysis 2: Comparison: Denosumab 180 mg vs Placebo; Test type: Superiority or Other; p = 0.133, van Elteren Stratified Rank Test

26. Secondary Outcome: Number of Participants With Anti-Denosumab Binding Antibodies
Description: Serum from participants was tested for antibodies to denosumab by immuoassay at months 1, 3, 6 and 12. The number of participants with anti-denosumab antibodies at any assessment is reported.
Time Frame: Assessed at Baseline and at Months 1, 3, 6 and 12.
Population: Patients who received at least 1 dose of investigational product and with at least one postbaseline sample taken.
Measure: Number; unit: Participants
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 72 | 70 | 75
Participants | 4 | 0 | 2

27. Secondary Outcome: Number of Participants With Anti-Denosumab Binding Antibody and Neutralizing Antibody
Description: Serum from participants testing positive for anti-denosumab binding antibodies was tested in a cell-based bioassay for neutralizing activity against denosumab.
Time Frame: Baseline to Month 12
Population: Patients who were positive for anti-denosumab antibodies
Measure: Number; unit: Participants
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 4 | 0 | 2
Participants | 0 |  | 0

28. Secondary Outcome: Change From Baseline in Albumin at Month 1
Description: Laboratory Chemistry Albumin
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 68 | 71
g/L | -0.36 (2.29) | -0.24 (2.25) | -0.30 (2.21)

29. Secondary Outcome: Change From Baseline in Albumin at Month 3
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 71
g/L | -0.30 (2.18) | -0.12 (2.28) | -0.18 (2.07)

30. Secondary Outcome: Change From Baseline in Albumin at Month 6
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 68 | 69
g/L | -0.30 (2.49) | -0.90 (2.56) | -0.77 (2.40)

31. Secondary Outcome: Change From Baseline in Albumin at Month 12
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 63
g/L | -0.13 (2.41) | -0.06 (2.26) | -0.59 (2.49)

32. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Month 1
Description: Laboratory chemistry alkaline phoshatatse
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
U/L | -5.87 (10.52) | -3.66 (11.97) | 1.18 (15.62)

33. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Month 3
Description: Laboratory chemisrty alkaline phosphatase
Time Frame: baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
U/L | -13.27 (15.91) | -12.38 (13.09) | -2.03 (8.37)

34. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Month 6
Description: Laboratory chemistry alkaline phosphatase
Time Frame: baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
U/L | -7.84 (31.94) | -12.49 (12.61) | -0.54 (18.46)

35. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Month 12
Description: Laboratory chemistry alkaline phosphatase
Time Frame: baseine, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
U/L | -11.92 (16.74) | -11.34 (18.18) | -4.63 (16.70)

36. Secondary Outcome: Change From Baseline in Bicarbonate at Month 1
Description: Laboratory chemistry bicarbonate
Time Frame: baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 67 | 70
mmol/L | 0.78 (2.31) | 0.06 (3.06) | 0.54 (2.94)

37. Secondary Outcome: Change From Baseline in Bicarbonate at Month 3
Description: Laboratory chemistry bicarbonate
Time Frame: baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 67 | 70
mmol/L | 0.12 (2.40) | 0.39 (2.84) | -0.67 (3.17)

38. Secondary Outcome: Change From Baseline in Bicarbonate at Month 6
Description: Laboratory chemistry bicarbonate
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 67 | 66
mmol/L | 0.45 (2.29) | -0.12 (2.61) | -0.18 (2.67)

39. Secondary Outcome: Change From Baseline in Bicarbonate at Month 12
Description: Laboratory chemistry bicarbonate
Time Frame: Baseline, Month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 62
mmol/L | 0.81 (2.12) | 0.58 (2.68) | 0.23 (2.50)

40. Secondary Outcome: Change From Baseline in Total Bilirubin at Month 1
Description: Laboratory chemistry total bilirubin
Time Frame: baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 67 | 70
umol/L | 0.26 (2.39) | -0.23 (2.45) | 0.42 (2.83)

41. Secondary Outcome: Change From Baseline in Total Bilirubin at Month 3
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 67 | 70
umol/L | 0.92 (2.17) | -0.23 (2.36) | 0.44 (2.74)

42. Secondary Outcome: Change From Baseline in Total Bilirubin at Month 6
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 67 | 66
umol/L | 1.08 (2.58) | -0.61 (2.49) | 0.34 (3.30)

43. Secondary Outcome: Change From Baseline in Total Bilirubin at Month 12
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 62
umol/L | 0.41 (2.58) | -0.35 (2.28) | 0.03 (2.80)

44. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen at Month 1
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
mmol/L | 0 (1.35) | 0.15 (1.40) | -0.01 (1.55)

45. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen at Month 3
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
mmol/L | 0.04 (1.35) | 0.41 (1.59) | 0.06 (1.43)

46. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen at Month 6
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
mmol/L | -0.21 (1.44) | -0.08 (1.41) | -0.04 (2.29)

47. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen at Month 12
Description: Laboratory chemistry blood urea nitrogen
Time Frame: baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
mmol/L | 0.32 (1.37) | 0.24 (1.46) | -0.09 (1.56)

48. Secondary Outcome: Change From Baseline in Calcium at Month 1
Description: Laboratory chemistry calcium
Time Frame: baseline. month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
mmol/L | -0.05 (0.11) | -0.05 (0.09) | 0.01 (0.09)

49. Secondary Outcome: Change From Baseline in Calcium at Month 3
Description: Laboratory chemistry calcium
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
mmol/L | -0.01 (0.11) | -0.02 (0.10) | 0 (0.10)

50. Secondary Outcome: Change From Baseline in Calcium at Month 6
Description: Laboratory chemistry calcium
Time Frame: baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
mmol/L | -0.01 (0.10) | -0.03 (0.11) | -0.01 (0.10)

51. Secondary Outcome: Change From Baseline in Calcium at Month 12
Description: Laboratory chemistry calcium
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
mmol/L | -0.01 (0.11) | 0.01 (0.09) | 0.01 (0.08)

52. Secondary Outcome: Change From Baseline in Calcium (Corrected) at Month 1
Description: Laboratory chemistry albumin-adjusted calcium
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
mmol/L | -0.05 (0.11) | -0.05 (0.09) | 0.01 (0.09)

53. Secondary Outcome: Change From Baseline in Calcium (Corrected) at Month 3
Description: Laboratory chemistry albumin-adjusted calcium
Time Frame: baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
mmol/L | -0.01 (0.11) | -0.02 (0.09) | 0 (0.10)

54. Secondary Outcome: Change From Baseline in Calcium (Corrected) at Month 6
Description: Laboratory chemistry albumin-adjusted calcium
Time Frame: Baseline, Month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
mmol/L | -0.01 (0.10) | -0.02 (0.10) | -0.01 (0.09)

55. Secondary Outcome: Change From Baseline in Calcium (Corrected) at Month 12
Description: Laboratory chemistry albumin-adjusted calcium
Time Frame: Baselien, Month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
mmol/L | -0.01 (0.11) | 0.01 (0.09) | 0 (0.08)

56. Secondary Outcome: Change From Baseline in Chloride at Month 1
Description: Laboratory chemistry chloride
Time Frame: baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 72
mmol/L | 0.24 (2.36) | 0.58 (2.66) | 0.01 (2.09)

57. Secondary Outcome: Change From Baseline in Chloride at Month 3
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 69 | 72
mmol/L | -0.01 (2.67) | 0.38 (2.35) | 0.78 (2.20)

58. Secondary Outcome: Change From Baseline in Chloride at Month 6
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 70
mmol/L | -0.57 (2.85) | 0.48 (2.19) | 0 (2.79)

59. Secondary Outcome: Change From Baseline in Chloride at Month 12
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 66 | 64
mmol/L | -0.62 (2.45) | -0.21 (2.58) | -0.08 (2.39)

60. Secondary Outcome: Change From Baseline in Creatinine at Month 1
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 72
µmol/L | -0.88 (9.89) | 0.38 (8.63) | 1.47 (8.78)

61. Secondary Outcome: Change From Baseline in Creatinine at Month 3
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 69 | 72
µmol/L | 0.62 (11.11) | 3.20 (8.30) | 3.81 (9.24)

62. Secondary Outcome: Change From Baseline in Creatinine at Month 6
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 70
µmol/L | 3.30 (10.97) | 3.84 (9.88) | 3.54 (11.60)

63. Secondary Outcome: Change From Baseline in Creatinine at Month 12
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 66 | 64
µmol/L | 5.44 (10.09) | 4.42 (9.59) | 3.73 (7.84)

64. Secondary Outcome: Change From Baseline in Gamma-Glutamyl Transferase at Month 1
Description: Laboratory chemistry gamma-glutamyl transferase
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
U/L | 1.04 (8.13) | -1.25 (9.67) | 0.26 (10.63)

65. Secondary Outcome: Change From Baseline in Gamma-Glutamyl Transferase at Month 3
Description: Laboratory chemistry gamma-glutamyl transferase
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
U/L | 2.32 (10.94) | 0.04 (9.90) | 1.51 (15.87)

66. Secondary Outcome: Change From Baseline in Gamma-Glutamyl Transferase at Month 6
Description: Laboratory chemistry gamma-glutamyl transferase
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
U/L | 7.37 (36.42) | 0.28 (12.70) | 5.67 (37.98)

67. Secondary Outcome: Change From Baseline in Gamma-Glutamyl Transferase at Month 12
Description: Laboratory chemistry gamma-glutamyl transferase
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
U/L | 2.98 (10.94) | 1.08 (16.09) | -1.38 (14.70)

68. Secondary Outcome: Change From Baseline in Glucose at Month 1
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 68 | 71
mmol/L | 0.06 (0.76) | 0.20 (0.65) | 0.05 (1.28)

69. Secondary Outcome: Change From Baseline in Glucose at Month 3
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 71
mmol/L | 0.08 (0.87) | 0.20 (0.63) | 0.04 (1.26)

70. Secondary Outcome: Change From Baseline in Glucose at Month 6
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 68 | 69
mmol/L | 0.12 (0.85) | 0.20 (0.65) | -0.05 (1.26)

71. Secondary Outcome: Change From Baseline in Glucose at Month 12
Description: Laboratory chemistry glucose
Time Frame: baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 63
mmol/L | -0.04 (0.66) | 0.22 (0.96) | 0.19 (1.27)

72. Secondary Outcome: Change From Baseline in Potassium at Month 1
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 72
mmol/L | 0.06 (0.38) | 0.06 (0.36) | 0.04 (0.36)

73. Secondary Outcome: Change From Baseline in Potassium at Month 3
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 69 | 72
mmol/L | -0.01 (0.39) | 0.06 (0.40) | 0.04 (0.38)

74. Secondary Outcome: Change From Baseline in Potassium at Month 6
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 70
mmol/L | 0.01 (0.44) | -0.01 (0.36) | 0 (0.42)

75. Secondary Outcome: Change From Baseline in Potassium at Month 12
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 66 | 64
mmol/L | -0.07 (0.44) | -0.08 (0.35) | -0.04 (0.43)

76. Secondary Outcome: Change From Baseline in Magnesium at Month 1
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 72
mmol/L | 0.01 (0.06) | 0.02 (0.06) | 0.01 (0.05)

77. Secondary Outcome: Change From Baseline in Magnesium at Month 3
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 68 | 72
mmol/L | -0.01 (0.06) | 0.02 (0.06) | 0 (0.06)

78. Secondary Outcome: Change From Baseline in Magnesium at Month 6
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 68 | 70
mmol/L | 0 (0.06) | 0.01 (0.06) | 0.01 (0.07)

79. Secondary Outcome: Change From Baseline in Magnesium at Month 12
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 65 | 64
mmol/L | -0.01 (0.06) | -0.01 (0.07) | -0.01 (0.08)

80. Secondary Outcome: Change From Baseline in Sodium at Month 1
Description: Laboratory chemistry sodium
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 69 | 72
mmol/L | -0.03 (1.93) | -0.06 (2.62) | 0.33 (2.03)

81. Secondary Outcome: Change From Baseline in Sodium at Month 3
Description: Change From Baseline in Sodium at Month 3
Time Frame: Baseline, Month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 71 | 69 | 72
mmol/L | -0.14 (2.13) | -0.16 (2.29) | 0.39 (2.38)

82. Secondary Outcome: Change From Baseline in Sodium at Month 6
Description: Laboratory chemistry sodium
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 69 | 70
mmol/L | -0.12 (1.98) | -0.06 (1.75) | 0.03 (2.27)

83. Secondary Outcome: Change From Baseline in Sodium at Month 12
Description: Laboratory chemistry sodium
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 66 | 64
mmol/L | -0.25 (2.02) | -0.27 (2.75) | 0.33 (2.38)

84. Secondary Outcome: Change From Baseline in Phosphorus at Month 1
Description: Laboratory chemistry phosphorus
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 68 | 71
mmol/L | -0.09 (0.16) | -0.06 (0.19) | 0.02 (0.14)

85. Secondary Outcome: Change From Baseline in Phosphorus at Month 3
Description: Laboratory chemistry phosphorus
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 68 | 71
mmol/L | -0.03 (0.16) | -0.03 (0.18) | 0.01 (0.20)

86. Secondary Outcome: Change From Baseline in Phosphorus at Month 6
Description: Laboratory chemistry phosphorus
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 68 | 68
mmol/L | -0.05 (0.17) | -0.01 (0.18) | 0.03 (0.19)

87. Secondary Outcome: Change From Baseline in Phosphorus at Month 12
Description: Change From Baseline in Phosphorus at Month 12
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 65 | 63
mmol/L | -0.05 (0.17) | 0 (0.17) | 0 (0.16)

88. Secondary Outcome: Change From Baseline in Total Protein at Month 1
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 68 | 71
g/L | -0.46 (3.56) | -0.40 (3.22) | 0.21 (3.00)

89. Secondary Outcome: Change From Baseline in Total Protein at Month 3
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 71
g/L | -0.29 (3.35) | 0.07 (3.42) | -0.20 (3.54)

90. Secondary Outcome: Change From Baseline in Total Protein at Month 6
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 68 | 69
g/L | -0.09 (4.13) | -0.62 (3.40) | -0.57 (3.19)

91. Secondary Outcome: Change From Baseline in Total Protein at Month 12
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 63
g/L | -0.97 (3.76) | -0.91 (3.55) | -0.98 (3.10)

92. Secondary Outcome: Change From Baseline in Aspartate Amino Transferase at Month 1
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 68 | 71
U/L | -0.79 (5.84) | -0.26 (8.14) | 0.90 (8.35)

93. Secondary Outcome: Change From Baseline in Aspartate Amino Transferase at Month 3
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 68 | 71
U/L | 1.99 (5.77) | 0.40 (8.78) | 2.69 (9.37)

94. Secondary Outcome: Change From Baseline in Aspartate Amino Transferase
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 68 | 68
U/L | 3.85 (15.66) | 0.87 (7.58) | 3.24 (15.90)

95. Secondary Outcome: Change From Baseline in Aspartate Amino Transferase at Month 12
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 65 | 63
U/L | 3.86 (18.62) | 3.75 (18.11) | 2.24 (7.32)

96. Secondary Outcome: Change From Baseline in Alanine Amino Transferase at Month 1
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 67 | 70
U/L | -1.84 (8.61) | -1.03 (12.37) | 1.20 (15.44)

97. Secondary Outcome: Change From Baseline in Alanine Amino Transferase at Month 3
Description: Laboratory Chemistry alanine amino transferase
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 67 | 70
U/L | 0.04 (8.85) | -2.10 (14.34) | 1.54 (13.00)

98. Secondary Outcome: Change From Baseline in Alanine Amino Transferase at Month 6
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 65 | 67 | 66
U/L | 1.20 (15.83) | -1.76 (14.12) | 5.44 (51.19)

99. Secondary Outcome: Change From Baseline in Alanine Amino Transferase at Month 12
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 62
U/L | 4.86 (24.46) | 1.66 (14.30) | 1.82 (14.41)

100. Secondary Outcome: Change From Baseline in Basophils at Month 1
Description: Laboratory hematology basophils
Time Frame: baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: *10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 69
*10^9/L | 0 (0.07) | 0 (0.07) | -0.01 (0.07)

101. Secondary Outcome: Change From Baseline in Basophils at Month 3
Description: Laboratory hematology basophils
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 64 | 67
* 10^9/L | -0.01 (0.06) | -0.01 (0.07) | -0.01 (0.07)

102. Secondary Outcome: Change From Baseline in Basophils at Month 6
Description: Laboratory hematology basophils
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 66
* 10^9/L | 0 (0.06) | 0 (0.07) | 0 (0.06)

103. Secondary Outcome: Change From Baseline in Basophils at Month 12
Description: Laboratory hematology basophils
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 60
* 10^9/L | 0.02 (0.09) | 0 (0.09) | 0.03 (0.07)

104. Secondary Outcome: Change From Baseline in Eosinophils at Month 1
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 69
* 10^9/L | -0.02 (0.09) | -0.01 (0.09) | 0.01 (0.08)

105. Secondary Outcome: Change From Baseline in Eosinophils at Month 3
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 64 | 67
* 10^9/L | 0 (0.10) | 0 (0.10) | -0.01 (0.09)

106. Secondary Outcome: Change From Baseline in Eosinophils at Month 6
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 66
* 10^9/L | -0.03 (0.09) | 0 (0.13) | 0 (0.13)

107. Secondary Outcome: Change From Baseline in Eosinophils at Month 12
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 60
* 10^9/L | 0.03 (0.16) | 0.02 (0.12) | 0.01 (0.12)

108. Secondary Outcome: Change From Baseline in Hematocrit at Month 1
Description: Laboratory hematology hematocrit
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 70
Proportion of red blood cells in blood | 0 (0.02) | 0 (0.02) | 0 (0.02)

109. Secondary Outcome: Change From Baseline in Hematocrit at Month 3
Description: Laboratory hematology hematocrit
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 64 | 70
Proportion of red blood cells in blood | 0.01 (0.02) | 0 (0.03) | 0 (0.03)

110. Secondary Outcome: Change From Baseline in Hematocrit at Month 6
Description: Laboratory hematology hematocrit
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 67
Proportion of red blood cells in blood | 0.01 (0.02) | 0 (0.03) | 0 (0.03)

111. Secondary Outcome: Change From Baseline in Hematocrit at Month 12
Description: Laboratory hematology hematocrit
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 61
Proportion of red blood cells in blood | 0 (0.02) | 0 (0.03) | -0.01 (0.03)

112. Secondary Outcome: Change From Baseline in Hemoglobin at Month 1
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 70
g/L | -0.33 (6.73) | -1.48 (6.39) | -0.69 (6.34)

113. Secondary Outcome: Change From Baseline in Hemoglobin at Month 3
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 64 | 70
g/L | 0.69 (7.02) | -1.02 (8.36) | -1.10 (6.30)

114. Secondary Outcome: Change From Baseline in Hemoglobin at Month 6
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 67
g/L | -0.36 (7.80) | -1.69 (8.82) | -0.69 (8.21)

115. Secondary Outcome: Change From Baseline in Hemoglobin at Month 12
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 61
g/L | 1.21 (9.26) | 0.02 (11.66) | -0.46 (10.08)

116. Secondary Outcome: Change From Baseline in Lymphocytes at Month 1
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 69
* 10^9/L | -0.02 (0.41) | 0.10 (0.40) | 0 (0.45)

117. Secondary Outcome: Change From Baseline in Lymphocytes at Month 3
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 64 | 67
* 10^9/L | 0.07 (0.38) | 0.14 (0.48) | 0.08 (0.46)

118. Secondary Outcome: Change From Baseline in Lymphocytes at Month 6
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 66
* 10^9/L | 0.12 (0.41) | 0.05 (0.35) | 0.03 (0.68)

119. Secondary Outcome: Change From Baseline in Lymphocytes at Month 12
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 60
* 10^9/L | -0.02 (0.49) | 0.04 (0.50) | -0.02 (0.49)

120. Secondary Outcome: Change From Baseline in Monocytes at Month 1
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 69
* 10^9/L | 0.01 (0.13) | -0.01 (0.10) | 0.01 (0.12)

121. Secondary Outcome: Change From Baseline in Monocytes at Month 3
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 64 | 67
* 10^9/L | 0.02 (0.11) | 0.01 (0.11) | 0.02 (0.11)

122. Secondary Outcome: Change From Baseline in Monocytes at Month 6
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 66
* 10^9/L | 0.05 (0.17) | 0.04 (0.12) | 0.04 (0.13)

123. Secondary Outcome: Change From Baseline in Monocytes at Month 12
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 60
* 10^9/L | 0.03 (0.15) | 0 (0.11) | 0.02 (0.13)

124. Secondary Outcome: Change From Baseline in Total Neutrophils at Month 1
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 69
* 10^9/L | 0 (1.97) | 0.18 (1.99) | -0.13 (1.68)

125. Secondary Outcome: Change From Baseline in Total Neutrophils at Month 3
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 64 | 67
* 10^9/L | 0.11 (1.92) | 0.26 (1.64) | -0.11 (1.55)

126. Secondary Outcome: Change From Baseline in Total Neutrophils at Month 6
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 66
* 10^9/L | 0.18 (1.67) | -0.05 (1.66) | 0.27 (2.36)

127. Secondary Outcome: Change From Baseline in Total Neutrophils at Month 12
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 60
* 10^9/L | 0.65 (2.37) | 0.04 (1.79) | 0.10 (2.31)

128. Secondary Outcome: Change From Baseline in Platelets at Month 1
Description: Laboratory hematology platelets
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 64 | 68
* 10^9/L | 1.78 (44.53) | 10.36 (49.34) | 2.96 (44.15)

129. Secondary Outcome: Change From Baseline in Platelets at Month 3
Description: Laboratory hematology platelets
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 67 | 63 | 69
* 10^9/L | -2.82 (48.86) | 6.86 (50.18) | -1.97 (45.94)

130. Secondary Outcome: Change From Baseline in Platelets at Month 6
Description: Laboratory hematology platelets
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 62 | 65 | 65
* 10^9/L | 1.95 (54.95) | 1.00 (45.64) | 1.57 (53.39)

131. Secondary Outcome: Change From Baseline in Platelets at Month 12
Description: Laboratory hematology platelets
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 62 | 59
* 10^9/L | 3.32 (51.66) | -4.26 (51.12) | 1.07 (58.16)

132. Secondary Outcome: Change From Baseline in Red Blood Cells at Month 1
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 70
* 10^9/L | -0.01 (0.21) | -0.01 (0.20) | -0.01 (0.19)

133. Secondary Outcome: Change From Baseline in Red Blood Cells at Month 3
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 64 | 70
* 10^9/L | 0.05 (0.23) | 0.02 (0.28) | 0 (0.23)

134. Secondary Outcome: Change From Baseline in Red Blood Cells at Month 6
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 67
* 10^9/L | 0.01 (0.24) | -0.04 (0.26) | 0.01 (0.26)

135. Secondary Outcome: Change From Baseline in Red Blood Cells at Month 12
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 61
* 10^9/L | 0.01 (0.27) | -0.06 (0.30) | -0.03 (0.29)

136. Secondary Outcome: Change From Baseline in White Blood Cells at Month 1
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 1
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 1.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 66 | 64 | 70
* 10^9/L | -0.03 (2.07) | 0.26 (2.04) | -0.10 (1.88)

137. Secondary Outcome: Change From Baseline in White Blood Cells at Month 3
Description: Laboratpry hematology white blood cells
Time Frame: Baseline, month 3
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 64 | 70
* 10^9/L | 0.18 (1.93) | 0.40 (1.71) | -0.05 (1.64)

138. Secondary Outcome: Change From Baseline in White Blood Cells at Month 6
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 6
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 64 | 65 | 67
* 10^9/L | 0.30 (1.78) | 0.04 (1.85) | 0.35 (2.34)

139. Secondary Outcome: Change From Baseline in White Blood Cells at Month 12
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 12
Population: Subjects who received at least 1 dose of investigational product who had nonmissing data at baseline and month 12.
Measure: Mean (Standard Deviation); unit: * 10^9/L
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 61 | 62 | 61
* 10^9/L | 0.70 (2.40) | 0.11 (1.86) | 0.13 (2.22)

140. Secondary Outcome: Number of Participants With Laboratory Common Terminology Criteria for Adverse Events (CTCAE) Grade Greater or Equal to 3
Description: Participants with laboratory toxicity of grade 3 or 4, graded according to the Common Terminology Criteria for Adverse Events, version 3.0, on the following general guideline:
  Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death related to AE.
Time Frame: Month 1, month 3, month 6, month 12
Population: Patients who received at least 1 dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Denosumab 180 mg | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 72 | 71 | 75
Participants
  Alanine Amino Transferase-above normal (grade 3) | 0 | 0 | 1
  Aspartate Amino Transferase-above normal (grade 3) | 0 | 1 | 0
  Glucose-above normal (grade 3) | 1 | 0 | 0
  Lymphocytes-below normal (grade 3) | 1 | 3 | 2
  Sodium-below normal (grade 3) | 1 | 2 | 0
  White Blood Cells-below normal (grade 3) | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Denosumab 60 mg | Denosumab 180 mg
Serious Adverse Events (participants affected / at risk) | 5/75 | 3/71 | 6/72
Other Adverse Events (participants affected / at risk) | 47/75 | 44/71 | 44/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Denosumab 60 mg (N=71) | Denosumab 180 mg (N=72)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Denosumab 60 mg (N=71) | Denosumab 180 mg (N=72)
Fatigue (General disorders) | 3 | 6 | 0
Bronchitis (Infections and infestations) | 3 | 3 | 4
Influenza (Infections and infestations) | 0 | 2 | 6
Nasopharyngitis (Infections and infestations) | 9 | 5 | 5
Sinusitis (Infections and infestations) | 8 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 11 | 8
Urinary tract infection (Infections and infestations) | 1 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 24 | 22 | 21
Dizziness (Nervous system disorders) | 4 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 4 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.